CLINICAL TRIAL: NCT05548270
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Efficacy and Safety of DPI-386 Nasal Gel for the Prevention of Nausea and Vomiting Associated With Motion
Brief Title: Efficacy and Safety of DPI-386 Nasal Gel for the Prevention of Nausea and Vomiting Associated With Motion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPI-386-MS-33
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DPI-386 (Experimental): Each 0.12 gram of the gel contains0.2 mg of scopolamine HBr
  Interventions: Drug: DPI-386 Nasal Gel
- Placebo (Placebo Comparator): Placebo Nasal Gel (0.12 g)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — Subjects will self-administer DPI-386 Nasal Gel or Placebo
  Other Names: scopolamine
  Arms: DPI-386
Drug: Placebo — Subjects will self-administer DPI-386 Nasal Gel or Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled study evaluating DPI-386 Nasal Gel versus placebo. Approximately 500 subjects will be randomized 1:1 (250 DPI 386 Nasal Gel/250 matching Placebo Nasal Gel) are planned to be enrolled.

DETAILED DESCRIPTION:
The purpose of this study (DPI-386-MS-33) is to prospectively evaluate the difference in the rate of complete response, defined as no vomiting and no rescue treatment (e.g., antihistamine) within the 4-hour period after study drug administration, or to the end of the voyage, whichever comes later, between 0.2 mg scopolamine administered as the DPI-386 Nasal Gel and Placebo Nasal Gel to subjects ≥18 years of age (inclusive) with a history of symptoms consistent with motion sickness (MS). The sample size of 250 subjects per treatment arm is considered sufficient to demonstrate a statistically significant difference between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent prior to initiation of any study-related procedures, and ability in the opinion of the Investigator to understand and comply with all the requirements of the study, which includes abstaining from the use of prohibited medications.
2. Male and female subjects ≥18 years of age.
3. Susceptible to provocative motion as evidenced by at least three responses of "Frequently" from the Motion Sickness Susceptibility Questionnaire Short-Form (MSSQ-Short).
4. Acceptable overall medical condition to be safely enrolled in and complete the study in the opinion of the Investigator.
5. Ability to take intranasal medication.
6. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is 2 years postmenopausal), or females of child-bearing potential using an acceptable method of birth control (i.e., oral contraception, systemic [injectable or patch] contraception, double barrier methods, strict abstinence, condoms, diaphragm, spermicidal agents, cervical cap, copper intrauterine device, etc.) for a period of up to 30 days before dosing and for one month after dosing and must have a negative pregnancy test at screening.
7. Agree to adhere to the following lifestyle compliance considerations:

   1. Refrain from consumption of grapefruit and any substance containing grapefruit for 7 days prior to, during, and 7 days after study drug administration;
   2. Abstain from alcohol for 24 hours prior to the administration of study drug and throughout the ocean travel;
   3. Abstain from marijuana within the 7-day period prior to the Treatment Day and throughout Day 2.
8. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-COV-2) negative test, confirmed by Food and Drug Administration (FDA) authorized COVID-19 test ≤ 7 days prior to study drug administration or no COVID 19 symptoms 10 days prior to study drug administration.

Exclusion Criteria:

1. Nauseated prior to boarding.
2. Mini-Mental State Examination score of <24.
3. Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential, who:

   1. Are or intend to become pregnant (including use of fertility drugs) during the study;
   2. Are nursing (female subjects only);
   3. Are not using an acceptable, highly effective method of contraception until all follow up procedures are complete.
4. Known allergic reactions to scopolamine or other anticholinergics.
5. Hospitalization or significant surgery requiring hospital admittance within the past 6 months.
6. Treatment with another investigational product within the past 30 days.
7. Donated blood or plasma or suffered significant blood loss within the past 30 days.
8. Chronic nausea caused by conditions such as irritable bowel syndrome, gastroparesis, cyclic vomiting syndrome or any other cause.
9. Having any of the following medical conditions within the last 2 years or if any of the following medical conditions were experienced more than 2 years ago and are deemed as clinically significant by the Investigator:

   1. Significant gastrointestinal disorder, asthma, or seizure disorders;
   2. History of or current cardiovascular disease;
   3. History of or current vestibular disorders;
   4. History of or current narrow-angle glaucoma;
   5. History of or current urinary retention problems; or
   6. History of or current alcohol or drug abuse.
10. Has had any prior nasal, nasal sinus, or nasal mucosa surgery.
11. Currently taking any of the following medication types within the specified washout period:

    1. Any form of scopolamine (including Transderm Scop®/washout 5 days;
    2. Belladonna alkaloids/washout 14 days;
    3. Antihistamines (including meclizine/washout 14 days;
    4. Tricyclic antidepressants/washout 14 days;
    5. Muscle relaxants/washout 4 days; or
    6. Nasal decongestants/washout 4 days.
12. Has used marijuana within the 7-day period prior to the Treatment Day. (Note: this criterion will only be confirmed at Eligibility Confirmation, not at Recruitment and Screening, although heavy users of marijuana can be determined ineligible at Screening. All potential study subjects deemed eligible at Screening must be informed at that time that this requirement must be met at Eligibility Confirmation.).
13. Unwilling or unable to follow the medication restrictions or unwilling to wash-out the use of restricted medications as noted in Exclusion Criterion #11.
14. Subject participated in a previous study of DPI-386 Nasal Gel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Who Report no Vomiting Within 4 Hours or to end of voyage, whichever comes later after Receiving Study Drug and no Use of Rescue Treatment | 4 hours
  Proportion of subjects who report no vomiting within 4 hours or to end of voyage, whichever comes later, after receiving study drug and no use of rescue treatment (e.g., antihistamine) within 4 hours or to end of voyage, whichever comes later, after receiving study drug (Complete Responders).

SECONDARY OUTCOMES:
Time to vomiting or use of rescue medication | 4 hours
Proportion of subjects who did not have moderate or severe nausea, which is defined as those subjects who report no moderate and severe nausea within 4 hours after receiving study drug and who did not use rescue treatment | 4 hours
  Proportion of subjects who did not have moderate or severe nausea, which is defined as those subjects who report no moderate and severe nausea within 4 hours after receiving study drug and who did not use rescue treatment (e.g., antihistamine) within 4 hours after receiving study drug.
Proportion of subjects who did not have nausea, which is defined as those subjects who report no nausea within 4 hours after receiving study drug and who did not use rescue treatment | 4 hours
  Proportion of subjects who did not have nausea, which is defined as those subjects who report no nausea within 4 hours after receiving study drug and who did not use rescue treatment (e.g., antihistamine) within 4 hours after receiving study drug.

CONTACTS AND LOCATIONS:
Overall Officials: David Helton, Study Director — Defender Pharmaceuticals, Inc.
Locations (1):
- Santa Monica Clinical Trials, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No